CLINICAL TRIAL: NCT06525467
Title: Primary Renal Lymphoma: a Case Report and Review of the Literature.
Brief Title: Primary Renal Lymphoma on a 48 Year Old Woman
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Huber Díaz Fuentes, Dr., Instituto Mexicano del Seguro Social
Other Study IDs: 98255832
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Renal Lymphoma
Keywords: neoplasms, renal, primary
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: radical nephrectomy — open radical nephrectomy and lymph node dissection.

SUMMARY:
A 48-year-old female presented to our hospital with the following medical conditions: Systemic arterial hypertension in treatment. She denies any allergies or surgical history.

She reports a history of asthenia and adynamia for 3 months, accompanied by intermittent pain in the left flank. She denies hematuria, fever or weight loss. She underwent an enhanced CT examination at the local hospital, and a mass (10 x 9 cm in diameter) was noted in the left kidney.

DETAILED DESCRIPTION:
She underwent radical nephrectomy and lymph node dissection. with the following surgical findings: (Figure 3) Kidney measuring 7 x 6 x 5 cm, with a tumor located in the upper pole of approximately 12 cm, with abundant newly formed vessels, loose and firm adhesions tumor-spleen and tail of pancreas, 1 artery, 1 vein, 1 ureter.

Postoperative pathology and inmunohistochemistry indicated DLBCL wich only localized in the kidney. Bone marrow biopsy and CT of the chest region dod not show any evidence of linmphoma invasion. According to the findings, she was diagnosed with PRL. After operation the patient received the R-CHOP regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patient with renal lymphoma

Exclusion Criteria:

* Patient without renal lymphoma

Ages: 48 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 48 Year old female
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-06-22 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2024-06-22 (Actual)

PRIMARY OUTCOMES:
Cure of the disease | 5 days
  Complete cancer resection

CONTACTS AND LOCATIONS:
Locations (1):
- Mexican Institute Of Social Health, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: Yes
manuscript publication
Supporting Information: CSR
Time Frame: September for ever

REFERENCES:
- See also: Related Info — http://www.spandidos-publications.com/10.3892/ol.2016.5173